CLINICAL TRIAL: NCT01532687
Title: A Randomized, Double-Blind Phase II, Study of Gemcitabine Alone or in Combination With Pazopanib for Refractory Soft Tissue Sarcoma
Brief Title: Gemcitabine With or Without Pazopanib in Treating Patients With Refractory Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Christopher Ryan, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00007943; NCI-2012-00052 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB00007943 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2012-02-06; First posted 2012-02-14 (Estimated); Results first posted 2021-02-09 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Adult Alveolar Soft Part Sarcoma; Adult Angiosarcoma; Adult Desmoplastic Small Round Cell Tumor; Adult Epithelioid Hemangioendothelioma; Adult Epithelioid Sarcoma; Adult Extraskeletal Myxoid Chondrosarcoma; Adult Extraskeletal Osteosarcoma; Adult Fibrosarcoma; Adult Leiomyosarcoma; Adult Liposarcoma; Adult Malignant Peripheral Nerve Sheath Tumor; Adult Rhabdomyosarcoma; Adult Synovial Sarcoma; Adult Undifferentiated Pleomorphic Sarcoma; Malignant Adult Hemangiopericytoma; Recurrent Adult Soft Tissue Sarcoma; Sarcoma; Stage III Adult Soft Tissue Sarcoma AJCC v7; Stage IV Adult Soft Tissue Sarcoma AJCC v7
MeSH Terms: conditions — Sarcoma, Alveolar Soft Part; Hemangiosarcoma; Desmoplastic Small Round Cell Tumor; Hemangioendothelioma, Epithelioid; Sarcoma; Chondrosarcoma, Extraskeletal Myxoid; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Neurofibrosarcoma; Rhabdomyosarcoma; Sarcoma, Synovial; Histiocytoma, Malignant Fibrous | interventions — Gemcitabine; pazopanib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (gemcitabine hydrochloride and pazopanib hydrochloride) (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and pazopanib hydrochloride PO on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Pazopanib; Drug: Pazopanib Hydrochloride
- Arm II (gemcitabine hydrochloride, placebo) (Active Comparator): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and placebo PO on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression may receive single-agent pazopanib hydrochloride PO daily. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Pazopanib; Drug: Pazopanib Hydrochloride; Other: Placebo Administration

INTERVENTIONS:
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; FF 10832; FF-10832; FF10832; Gemcitabine HCI; Gemzar; LY-188011; LY188011
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pazopanib — Given PO
  Other Names: GW786034
Drug: Pazopanib Hydrochloride — Given PO
  Other Names: GW786034B; Votrient
Other: Placebo Administration — Given PO
  Arms: Arm II (gemcitabine hydrochloride, placebo)

SUMMARY:
This randomized phase II trial studies how well gemcitabine hydrochloride works with or without pazopanib hydrochloride in treating patients with refractory soft tissue sarcoma. Drugs used in chemotherapy, such as gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Pazopanib hydrochloride may also stop the growth of tumor cells by blocking blood flow to the tumor. It is not yet known whether gemcitabine hydrochloride is more effective with or without pazopanib hydrochloride in treating patients with soft tissue sarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate whether treatment with gemcitabine (gemcitabine hydrochloride) plus pazopanib (pazopanib hydrochloride) improves the median progression-free survival (PFS) of patients with metastatic soft tissue sarcoma when compared to gemcitabine plus placebo.

SECONDARY OBJECTIVES:

I. To assess overall response in this population to gemcitabine plus pazopanib compared to gemcitabine plus placebo.

II. To assess overall survival (OS) in this population to gemcitabine plus pazopanib compared to gemcitabine plus placebo.

III. To investigate differences in treatment response in different histologic subgroups (liposarcoma vs. all other eligible soft tissue sarcoma subtypes).

IV. To evaluate the safety and tolerability of the combination of gemcitabine plus pazopanib.

V. To assess the progression-free survival and overall response in patients treated with single agent pazopanib following administration of gemcitabine in the cross-over portion of this study.

VI. To collect specimens for an exploratory analysis of potential biomarkers that predict response in patients receiving combination therapy with gemcitabine plus pazopanib.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive gemcitabine hydrochloride intravenously (IV) over 30 minutes on days 1 and 8 and pazopanib hydrochloride orally (PO) on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and placebo PO on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression may receive single-agent pazopanib hydrochloride PO daily. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After the completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow-up; procedures conducted as part of the subject's routine clinical management (e.g., blood count, imaging study) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol
* Histologically confirmed diagnosis of metastatic or unresectable soft tissue sarcoma, excluding gastrointestinal stromal tumors, Kaposi's sarcoma, Ewing's family of tumors, and embryonal or alveolar rhabdomyosarcoma
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Patients must have received at least one, but not more than three, systemic regimens for treatment of metastatic soft tissue sarcoma; patients must have had a prior anthracycline in the neoadjuvant, adjuvant, or metastatic setting unless medically inappropriate for the patient
* Neoadjuvant or adjuvant therapy will not count towards prior treatment for metastatic disease, unless the patient relapsed within 2 years of completing such therapy.
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Hemoglobin >= 8 g/dL; subjects may not have had a transfusion within 7 days of screening assessment
* Platelets >= 100 x 10^9/L
* Prothrombin time (PT) or international normalized ratio (INR) =< 1.2 x upper limit of normal (ULN); subjects receiving anticoagulation therapy are eligible if their INR is stable and within the recommended range for the desired level of anticoagulation
* Activated partial thromboplastin time (aPTT) =< 1.2 x ULN
* Total bilirubin =< 1.5 x ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN; concomitant elevations in bilirubin and AST/ALT above 1.0 x ULN (upper limit of normal) are not permitted
* Serum creatinine =< 1.5 mg/dL (133 umol/L)
* Or, if > 1.5 mg/dL: calculated creatinine clearance (ClCR) >= 30 mL/min
* Urine protein to creatinine ratio (UPC) < 1; if UPC >= 1, then a 24-hour urine protein must be assessed; subjects must have a 24-hour urine protein value < 1 g to be eligible; use of urine dipstick for renal function assessment is not acceptable
* Or 24-hour urine protein < 1 g
* A female is eligible to enter and participate in this study if she is of:

  * Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had:

    * A hysterectomy
    * A bilateral oophorectomy (ovariectomy)
    * A bilateral tubal ligation
    * Is post-menopausal
* Subjects not using hormone replacement therapy (HRT) must have experienced total cessation of menses for >= 1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone (FSH) value > 40 mIU/mL and an estradiol value < 40 pg/mL (< 140 pmol/L)
* Subjects using HRT must have experienced total cessation of menses for >= 1 year and be greater than 45 years of age OR have had documented evidence of menopause based on FSH and estradiol concentrations prior to initiation of HRT
* Childbearing potential, including any female who has had a negative serum pregnancy test within 7 days prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception; defined as follows:

  * Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product
  * Oral contraceptive, either combined or progesterone alone
  * Injectable progesterone
  * Implants of levonorgestrel
  * Estrogenic vaginal ring
  * Percutaneous contraceptive patches
  * Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year
  * Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject
  * Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository)
* Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug

Exclusion Criteria:

* Prior malignancy; note: subjects who have had another malignancy and have been disease-free for > 3 years, or subjects with a history of completely resected non-melanomatous skin carcinoma, successfully treated in situ carcinoma, or successfully treated superficial bladder cancer are eligible.
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 months prior to first dose of study drug; screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required only if clinically indicated or if the subject has a history of CNS metastases
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

  * Active peptic ulcer disease
  * Known intraluminal metastatic lesion/s with risk of bleeding
  * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

  * Malabsorption syndrome
  * Major resection of the stomach or small bowel
* Presence of uncontrolled infection
* Corrected QT interval (QTc) > 480 msecs using Bazett's formula
* History of any one or more of the following cardiovascular conditions within the past 6 months:

  * Cardiac angioplasty or stenting
  * Myocardial infarction
  * Unstable angina
  * Coronary artery bypass graft surgery
  * Symptomatic peripheral vascular disease
* Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
* Poorly controlled hypertension (defined as systolic blood pressure [SBP] of >= 140 mmHg or diastolic blood pressure [DBP] of >= 90mmHg); note: initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry; following antihypertensive medication initiation or adjustment, blood pressure (BP) must be re-assessed three times at approximately 2-minute intervals; at least 24 hours must have elapsed between anti-hypertensive medication initiation or adjustment and BP measurement; these three values should be averaged to obtain the mean diastolic blood pressure and the mean systolic blood pressure; the mean SBP/DBP ratio must be < 140/90 mmHg
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months; note: subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major)
* Evidence of active bleeding or bleeding diathesis
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage
* Hemoptysis in excess of 2.5 mL (or one half teaspoon) within 8 weeks of first dose of study drug
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures
* Unable or unwilling to discontinue use of prohibited medications for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study; administration of any non-oncologic investigational drug within 30 days or 5 half-lives whichever is longer prior to receiving the first dose of study treatment
* Treatment with any of the following anti-cancer therapies:

  * Radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib OR
  * Chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days (or 28 days in the case of monoclonal antibody therapy) prior to the first dose of pazopanib.
  * Any prior treatment with pazopanib.
  * Prior treatment with vascular endothelial growth factor (VEGF) or vascular endothelial growth factor receptor (VEGFR)-targeting agents other than pazopanib (eg. sorafenib, sunitinib, and bevacizumab) in the metastatic setting. Prior use of such agents in the neoadjuvant or adjuvant setting is permitted.
  * Any prior treatment with gemcitabine for metastatic disease. Prior use of gemcitabine in the neoadjuvant or adjuvant setting is permitted.
* Any ongoing toxicity from prior anti-cancer therapy that is > grade 1 and/or that is progressing in severity, except alopecia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-03-13 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W Ryan, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Double-blinded randomization (1:1) was stratified by subtypes of sarcoma (liposarcoma vs. all other eligible soft tissue sarcoma subtypes). Patients were randomized to either experimental arm or placebo arm prior to starting treatment. Those who discontinued treatment on the placebo arm due to disease progression were eligible for treatment with open-label pazopanib (unblinded, cross-over treatment); those who developed disease progression on the Experimental arm (pazopanib arm) were not.
Groups:
- Gemcitabine Hydrochloride Plus Pazopanib Hydrochloride: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and pazopanib hydrochloride PO on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Gemcitabine: Given IV
  Gemcitabine Hydrochloride: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Pazopanib: Given PO
  Pazopanib Hydrochloride: Given PO
- Gemcitabine Hydrochloride Plus Placebo: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and placebo PO on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression may receive single-agent pazopanib hydrochloride PO daily. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Gemcitabine: Given IV
  Gemcitabine Hydrochloride: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Pazopanib: Given PO
  Pazopanib Hydrochloride: Given PO
  Placebo Administration: Given PO
Period: Overall Study
Arm/Group | Gemcitabine Hydrochloride Plus Pazopanib Hydrochloride | Gemcitabine Hydrochloride Plus Placebo
Started | 29 | 25
Crossover to Open-label Pazopanib (Participants who progress, unblinded, and found treated with gemcitibine+placebo arm are eligible to crossover into pazopanib open-label treatment phase) | 0 | 14
Completed | 15 (Participants remain on treatment until time of progression and through the AE assessment period) | 23 (Participants remain on treatment until time of progression)
Not Completed | 14 | 2
Not completed — Death | 2 | 0
Not completed — Adverse Event | 6 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 2 | 1
Not completed — Protocol-defined delay > 3 weeks | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcitabine Hydrochloride Plus Pazopanib Hydrochloride | Gemcitabine Hydrochloride Plus Placebo | Total
Number analyzed (Participants) | 29 | 25 | 54
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [55 to 70] | 56 [48 to 66] | 60 [50.3 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 15 | 9 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  White | 25 | 24 | 49
  Unknown/Not Reported | 3 | 1 | 4
Histology [Count of Participants; unit: Participants]
  Liposarcoma | 9 | 7 | 16
  Leiomyosarcoma (LMS) | 9 | 5 | 14
  Undifferentiated Pleomorphic Sarcoma (UPS) | 3 | 5 | 8
  Synovial Sarcoma | 3 | 3 | 6
  Other Sarcoma(s) | 5 | 5 | 10
Number Prior Treatments [Median (Full Range); unit: Treatments] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Compared using a one-sided Gehan-Wilcoxon test stratified by sarcoma subtype. Kaplan-Meier estimates for each treatment arm will be presented with the estimated hazard ratios and their associated confidence intervals. Progression is defined using Response Evaluation Criteria in Solid Tumors (RECIST) v1.0 as at least a 20% increase in the sum of the longest diameters of target lesions (taking as reference the smallest sum on study) with an absolute increase of at least 5 mm (target lesions), or measurable increase in non-target lesions (unequivocal progression), or appearance of one or more new lesions.
Time Frame: Calculated as the time from randomization to the first documented progression or death, whichever occurs first, or until time of last contact if no progression or death occurred, assessed up to 3 years
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine Hydrochloride Plus Pazopanib Hydrochloride | Gemcitabine Hydrochloride Plus Placebo
Number analyzed (Participants) | 29 | 25
months
  All randomized | 4.5 [3.0 to 8.5] | 1.6 [1.4 to 4.3]
  Liposarcoma: number analyzed (Participants) | 9 | 7
  Liposarcoma | 8.9 [4.3 to NA] — There were not sufficient events to define the upper limit of the confidence interval (two out of nine participants progressed) | 1.5 [1.0 to NA] — Due to the small sample size (n = 7) the upper confidence limit was not estimable (did not cross the 50% line)
  Other Sarcoma: number analyzed (Participants) | 20 | 18
  Other Sarcoma | 4.4 [3.0 to 8.8] | 2.2 [1.4 to 4.6]
Statistical Analysis 1: Comparison: Gemcitabine Hydrochloride Plus Pazopanib Hydrochloride vs Gemcitabine Hydrochloride Plus Placebo; Statistical results are for the full randomized population (n = 54). The study was originally designed with overall one-sided alpha of 5%, where a total of 73 patients (36 in the gemcitabine + placebo arm, and 37 in the gemcitabine + pazopanib arm) were required to achieve 80% power to detect a 2.5 month increase in median PFS (a hazard ratio of 0.55) between the two treatment arms. Study was closed early by the sponsor due to slow accrual and funds and thus was under powered; Test type: Superiority — Log-log plots revealed crossing of the curves at late time points, indicating a possible interaction between treatment arms over time. We used the Gehan-Wilcoxon test, which weights early differences between groups, to test whether there is a difference between the treatment arms early in the study; p = 0.017, Gehan-Wilcoxon
Statistical Analysis 2: Comparison: Gemcitabine Hydrochloride Plus Pazopanib Hydrochloride vs Gemcitabine Hydrochloride Plus Placebo; Comparison between the two arms for the liposarcoma subgroup; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.195, Gehan-Wilcoxon
Statistical Analysis 3: Comparison: Gemcitabine Hydrochloride Plus Pazopanib Hydrochloride vs Gemcitabine Hydrochloride Plus Placebo; Statistical results are for the 'other' sarcoma subgroup (n = 38); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.079, Gehan-Wilcoxon

2. Secondary Outcome: Progression-free Survival (PFS) for a Sub-group of Patients Treated With Open-label Pazopanib Hydrochloride Following Administration of Gemcitabine Hydrochloride in the Cross-over Portion of This Study
Description: Participants who progress during treatment and are found to be part of the gemcitabine+placebo arm after unblinding are eligible to receive open-label pazopanib with gemcitabine. This is the crossover population. Statistical analysis is exploratory and requires sufficient crossover participants to assess Kaplan-Meier estimated hazard ratio and associated 95% confidence interval. This represents the participants second progression. In both cases progression is defined using Response Evaluation Criteria in Solid Tumors (RECIST) v1.0 as at least a 20% increase in the sum of the longest diameters of target lesions with an absolute increase of at least 5 mm (target lesions), or measurable increase in non-target lesions (unequivocal progression), or appearance of one or more new lesions. First progression uses the smallest sum on study as a reference; progression for the crossover population uses first progression measurements as the reference.
Time Frame: Calculated as the time from receiving open-labeled pazopanib hydrochloride to the next documented progression or death whichever occurs first, assessed up to 3 years
Population: Participants randomized to the gemcitabine + placebo arm who progressed and elected to receive gemcitibine + open-label pazopanib
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Crossover From Gemcitabine + Placebo to Gemcitabine + Open-label Pazopanib: Participants randomized to the gemcitabine + placebo arm who progressed can be moved into the crossover arm, receiving gemcitabine + open-label pazopanib
Arm/Group | Crossover From Gemcitabine + Placebo to Gemcitabine + Open-label Pazopanib
Number analyzed (Participants) | 14
months | 3.0 [1.3 to NA] — Due to the small sample size (n = 14) the upper confidence limit was not estimable (did not cross the 50% line)

3. Secondary Outcome: Percentage of Participants Achieving Best Overall Objective Response (CR+PR)
Description: Response is evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, where RECIST combines assessments for target, non-target and presence of new lesions. Best Overall Objective Response is the sum of all CR+PR divided by all randomized participants, where the strongest recorded response is used for the evaluation (CR>PR>SD>PD). Objective response (CR+PR) requires at least a 30% decrease in the sum of the largest diameter target lesions (with respective to the baseline sum); disappearance of all or persistence of one or more non-target lesions, maintenance of tumor marker levels above normal limits, and no new lesions. Estimated odds ratio of best overall objective response are reported with 95% confidence interval for the two histologic sarcoma subgroups (liposarcoma vs all other eligible soft tissue sarcoma subtypes). One-sided proportions test is used to determine whether best overall objective response is greater for the gemcitabine plus pazopanib group.
Time Frame: Best overall objective response recorded from the start of treatment until disease progression/recurrence assessed up to 3 years
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine Hydrochloride Plus Pazopanib Hydrochloride | Gemcitabine Hydrochloride Plus Placebo
Number analyzed (Participants) | 29 | 25
percentage of participants
  All randomized participants | 6.9 [0.9 to 22.8] | 8.0 [1.0 to 26.0]
  Liposarcoma participants: number analyzed (Participants) | 9 | 7
  Liposarcoma participants | 22.2 [2.8 to 60] | 0 [NA to NA] — No participants achieved overall objective response, making the confidence interval not estimable
  Other sarcoma participants: number analyzed (Participants) | 20 | 18
  Other sarcoma participants | 0 [NA to NA] — No participants achieved overall objective response, making the confidence interval not estimable | 11.1 [1.4 to 34.7]
Statistical Analysis 1: Comparison: Gemcitabine Hydrochloride Plus Pazopanib Hydrochloride vs Gemcitabine Hydrochloride Plus Placebo; Statistical results are for the full randomized population (n = 54). The study tests whether gemcitabine plus pazopanib is superior to gemcitabine plus placebo (one-sided proportion test with Yate's continuity correction); Test type: Superiority — Analysis was not powered for secondary endpoints. Given the study closed early due to slow enrollment, we do not anticipate detecting a statistical difference between the two groups; p = 0.5, One-sided Proportions Test — Yate's continuity correction was applied because of the number of subjects and successes (n = 4)
Statistical Analysis 2: Comparison: Gemcitabine Hydrochloride Plus Pazopanib Hydrochloride vs Gemcitabine Hydrochloride Plus Placebo; Statistical results are for the Liposarcoma group (n = 16). The study tests whether gemcitabine plus pazopanib is superior to gemcitabine plus placebo (one-sided proportion test with Yate's continuity correction). Analysis was not powered for the secondary endpoints. Given the study closed early due to slow enrollment we do not anticipate detecting a statistical difference between the groups; Test type: Superiority; p = 0.3, One-sided Proportion Test — Yate's continuity correction was applied because of small number of participants (n = 16) and successes (n = 2)
Statistical Analysis 3: Comparison: Gemcitabine Hydrochloride Plus Pazopanib Hydrochloride vs Gemcitabine Hydrochloride Plus Placebo; Statistical results are for the Other Sarcoma group (n = 38). The study tests whether gemcitabine plus pazopanib is superior to gemcitabine plus placebo (one-sided proportion test with Yate's continuity correction). Analysis was not powered for secondary endpoints. Given the study closed early due to slow enrollment, we do not anticipate detecting a statistical difference between the two groups; Test type: Superiority; p = 0.8, One-sided Proportion Test — Yate's continuity correction was applied because of the small number of participants and successes (n = 2)

4. Secondary Outcome: Overall Survival
Description: Two treatment arms will be compared using a one-sided log-rank test stratified by sarcoma subtype and study site. Kaplan-Meier estimates and the survival curves for each treatment arm will be presented with the estimated hazard ratios and their associated confidence interval.
Time Frame: From randomization to death due to any cause, or until last patient contact if the patient did not die, assessed up to 3 years
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine Hydrochloride Plus Pazopanib Hydrochloride | Gemcitabine Hydrochloride Plus Placebo
Number analyzed (Participants) | 29 | 25
months
  All Randomized | 11.0 [9.6 to 20.7] | 15.6 [6.1 to 27.0]
  Liposarcoma participants: number analyzed (Participants) | 9 | 7
  Liposarcoma participants | 20.5 [11.0 to NA] — Upper limit was not estimable because there was no observed death time greater than the median survival that touched or crossed -1,96 using the log-transformation of the survival function (ref: Formula 4.5.5, Klein JP and Moeschberger ML, Survival Analysis: Techniques for censored and truncated data). This is likely due to small sample size (n = 9). | 5.7 [3.5 to NA] — Upper limit was not estimable due to small sample size (n = 7) and failure to cross the 25% line.
  Other Sarcoma participants: number analyzed (Participants) | 20 | 18
  Other Sarcoma participants | 10.2 [7.6 to 20.7] | 17.7 [7.6 to 30.7]
Statistical Analysis 1: Comparison: Gemcitabine Hydrochloride Plus Pazopanib Hydrochloride vs Gemcitabine Hydrochloride Plus Placebo; Overall survival estimated among all randomized participants (n = 54); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.481, Gehan-Wilcoxon
Statistical Analysis 2: Comparison: Gemcitabine Hydrochloride Plus Pazopanib Hydrochloride vs Gemcitabine Hydrochloride Plus Placebo; Overall survival compared between the two arms for the liposarcoma subgroup (n = 16); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.353, Gehan-Wilcoxon
Statistical Analysis 3: Comparison: Gemcitabine Hydrochloride Plus Pazopanib Hydrochloride vs Gemcitabine Hydrochloride Plus Placebo; Overall survival comparison between the two treatment arms for the other sarcoma group (n = 38); Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.408, Gehan-Wilcoxon

ADVERSE EVENTS:
Time Frame: Adverse events were collected up 30 days after the last dose of study drugs while participant was in that Arm/Group. All-Cause Mortality was assessed up to 3 years. For SAEs and OAEs, the Gem+Pazo group was assessed up to 32.1 months; Gem+Placebo participants were assessed up to 36.0 months (30 days after progression). If Gem+Placebo participants crossed over to open-label Pazo after progression, any additional AEs were collected under the crossover arm (up to 16.6 months).
Description: All Serious Adverse Events (SAEs) are reported, irrespective of grade or attribution. For other Adverse Events (AEs), only those grade 3 or higher are collected with a threshold set at 3.5% within any arm. AEs and SAEs are assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Assessments are made by laboratory tests, physical exam, and other clinical measurements (e.g. ECGs, radiological scans, vital signs, etc.)
Groups:
- Gemcitabine Hydrochloride Plus Placebo: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and placebo PO on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression, are unblinded and found randomized to placebo arm may crossover to receive open-label pazopanib hydrochloride PO daily.
  AEs and deaths reported only while participant is in placebo arm/group.
  Gemcitabine: Given IV
  Gemcitabine Hydrochloride: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Pazopanib: Given PO
  Pazopanib Hydrochloride: Given PO
  Placebo Administration: Given PO
- Crossover From Gemcitabine Plus Placebo to Gemcitabine Plus Open-label Pazopanib: Patients who progress and found randomized to the placebo arm after unblinding are eligible for receipt of open-label gemcitabine plus pazopanib. Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and pazopanib hydrochloride PO on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. AEs and deaths collected during this treatment period
Arm/Group | Gemcitabine Hydrochloride Plus Pazopanib Hydrochloride | Gemcitabine Hydrochloride Plus Placebo | Crossover From Gemcitabine Plus Placebo to Gemcitabine Plus Open-label Pazopanib
All-Cause Mortality (participants affected / at risk) | 23/29 | 10/11 | 11/14
Serious Adverse Events (participants affected / at risk) | 8/29 | 6/25 | 5/14
Other Adverse Events (participants affected / at risk) | 25/29 | 14/25 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine Hydrochloride Plus Pazopanib Hydrochloride (N=29) | Gemcitabine Hydrochloride Plus Placebo (N=25) | Crossover From Gemcitabine Plus Placebo to Gemcitabine Plus Open-label Pazopanib (N=14)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 1
Heart failure (Cardiac disorders) | 2 | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 2 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 1 | 0
Cardiac troponin I increase (Investigations) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Fever (General disorders) | 1 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Edema limbs (General disorders) | 1 | 0 | 0
Edema trunk (General disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine Hydrochloride Plus Pazopanib Hydrochloride (N=29) | Gemcitabine Hydrochloride Plus Placebo (N=25) | Crossover From Gemcitabine Plus Placebo to Gemcitabine Plus Open-label Pazopanib (N=14)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2
Alanine aminotransferase increased (Investigations) | 3 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 0
Heart failure (Cardiac disorders) | 2 | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 5 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Lymphocyte count decreased (Investigations) | 4 | 0 | 0
Neutrophil count decreased (Investigations) | 12 | 9 | 1
Platelet count decreased (Investigations) | 4 | 0 | 0
Thromboembolic event (Vascular disorders) | 3 | 0 | 0
White blood cell decreased (Investigations) | 4 | 1 | 0
Ejection fraction decreased (Investigations) | 2 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT01532687/Prot_SAP_000.pdf